CLINICAL TRIAL: NCT03951532
Title: Morbidity and Mortality Associated With the Care Journey in Children and Adolescents With Hyperthyroidism
Acronym: MOTHYRE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16010HLJ
Record Dates: First submitted 2019-03-12; First posted 2019-05-15 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2021-02

CONDITIONS: Hyperthyroidism
Keywords: Hyperthyroidism; paediatrics; health data base
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with hyperthyroidism: children and adolescents (6 months -17 years included) whose data are present in the SNIIRAM database (DCIR data) and beneficiaries of the general health insurance scheme during the study period (01/01/2006-31/12/2017)

SUMMARY:
"Early paediatric Basedow disease is one of the rare endocrine diseases for which the Reference Centre for Rare Endocrine Growth Diseases, was approved by the Ministry of Health in 2005. In addition, the study will benefit from the expertise of public Health France (SFP). This study is therefore part of the missions of these partners (reference centre for endocrine growth diseases and Public Health France).

For several years, our group has been interested in defining the evolutionary profile of these patients. A national study on short- and long-term patient follow-up has already been conducted, which has been the subject of two international publications29,30, as well as a study on a specific clinical form of the disease 24. This work was made possible thanks to the collaboration of paediatric clinical centres within the Reference Centre and Competence Centre for Rare Endocrine Diseases Network. The present study planned in France will make it possible to accurately characterize the care pathway and the frequency of complications associated with it at the national level.

DETAILED DESCRIPTION:
"With regard to the analysis of data on the identification of hyperthyroidism in children using the various medico-administrative databases, the epidemiological study of hyperthyroidism in children in France seems feasible using data on drug consumption from the SNIIRAM. These data will make it possible for the first time to study the impact of the disease in terms of serious morbidity and mortality (related to the disease and/or treatment) and to make recommendations for the management of the disease in order to improve the prognosis of the disease in children.

Thanks to these results, incidence data on the disease in children will be able to be estimated for the first time in France, as well as its temporal and spatial trends. They will be compared with national studies carried out in Sweden, Denmark and the United Kingdom on children. The spatial distribution in France can also be studied and compared with existing or emerging hypotheses, in particular concerning endocrine disrupters (French public health data). These analyses could also allow the generation of new causal hypotheses.

Finally, this work could lead to the establishment of national surveillance of hyperthyroidism in children. Prolonged follow-up is necessary, even after the end of medical treatment or after radical treatment, to determine the effectiveness of the management of patients during childhood and the impact on their overall health.

This study should therefore make it possible to propose recommendations to optimize the therapeutic management of hyperthyroidism in children and adolescents and improve the quality of life in adulthood for these patients.

The main objective of the study is to describe the complications (morbidity and mortality) associated with the 3 management modalities (treatment with synthetic antithyroid drugs (ATS), radioactive iodine and thyroidectomy) of children followed for hyperthyroidism in France, over a period of 11 years.

The study design chosen is that of an observational historical cohort study based on medico-administrative data from the National Inter-Regime Health Insurance Information System (SNIIRAM), which contains data from the PMSI (Information Systems Medicalization Program).

The study period begins on 01.01.2006 and ends on 31.12.2017.

ELIGIBILITY:
Inclusion Criteria:

* children from 6 months to 17 years old included,
* who received a dispensation of synthetic antithyroid drugs during the study period.

Exclusion Criteria:

* infants under 6 months of age,
* beneficiaries belonging to social security schemes other than the general scheme,
* children from multiple pregnancies.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes all children and adolescents (6 months -17 years included) whose data are present in the SNIIRAM database (DCIR data) and beneficiaries of the general health insurance scheme during the study period (01/01/2006-31/12/2017).
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
number of complications morbidity | for 11 years
  number of complications morbidity associated with the three management modalities (treatment with synthetic antithyroid drugs (ATS), radioactive iodine and thyroidectomy) of children followed for Maladie de Basedow in France, over a period of 11 years.
number of complications mortality | for 11 years
  number of complications morbidity associated with the three management modalities (treatment with synthetic antithyroid drugs (ATS), radioactive iodine and thyroidectomy) of children followed for Maladie de Basedow in France, over a period of 11 years.

SECONDARY OUTCOMES:
number of children and adolescents with a prescription or therapeutic modalities | for 11 years
  description of the therapeutic modalities of children and adolescents with Basedow's disease according to geographical distribution and time in France over a period of 11 years.
number of children with hyperthyroidism by geographical region and time in France | for 11 years
  Estimation of the prevalence and incidence of hyperthyroidism in children by geographical region and time in France over a period of 11 years
number of hyperthyroidism associated with other comorbidities | for 11 years
  Estimate of the number of hyperthyroidism associated with other co-morbidities, in particular cardiovascular disease, psychiatric disorders and cancer, in children according to geographical region and time in France over a period of 11 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Le Moal J, Chesneau J, Goria S, Boizeau P, Haignere J, Kaguelidou F, Leger J. Spatiotemporal variation of childhood hyperthyroidism: a 10-year nationwide study. Eur J Endocrinol. 2022 Oct 3;187(5):675-683. doi: 10.1530/EJE-22-0355. Print 2022 Nov 1. PMID 36074933